CLINICAL TRIAL: NCT01735188
Title: A Natural History Study Of Molybdenum Cofactor And Isolated Sulfite Oxidase Deficiencies
Status: Completed | Type: Observational
Sponsor: Origin Biosciences (Industry)
Responsible Party: Sponsor
Other Study IDs: ALX-MCD-502; ALX-MCD-502 (Registry Identifier: ALXN-MCD-502)
Record Dates: First submitted 2012-11-26; First posted 2012-11-28 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Molybdenum Cofactor Deficiency; Isolated Sulfite Oxidase Deficiency
Keywords: Natural history study
MeSH Terms: conditions — Molybdenum cofactor deficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Plasma, urine, whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Living
- Deceased

SUMMARY:
Primary objective:

Characterize the natural history of MoCD type A in terms of survival

Secondary objectives:

1. Evaluate blood and urine for biochemical markers
2. Evaluate head circumference, seizure activity and neurologic outcomes
3. To evaluate brain MRI
4. Compare blood and urine analysis, head circumference, seizure activity and neurologic outcomes to MRI findings

ELIGIBILITY:
Inclusion Criteria:

1. Both living and deceased patients of any age will be considered for study inclusion.
2. Diagnosis of MoCD or isolated SOX deficiency
3. Documented informed consent

Exclusion Criteria:

1. MoCD Type A patient who was in Study ALX-MCD-501
2. Deceased patients with unknown genotype (as of Amendment 4)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The actual sample size will depend on successful identification of at least 30 MoCD Type A patients
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2013-08; Primary Completion 2015-11 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
To characterize the natural history of molybdenum cofactor deficiency (MoCD) type A, the most common subtype of MoCD, in terms of survival | 12 months

SECONDARY OUTCOMES:
To evaluate levels of the biochemical markers S-sulfocysteine (SSC), uric acid, and xanthine in blood, urine, and cerebral spinal fluid over time in patients with MoCD and isolated sulfite oxidase (SOX) deficiency. | 12 months

CONTACTS AND LOCATIONS:
Locations (32):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - UVA Health System, Charlottesville, Virginia
  - Woodinville Pediatrics PLLC, Woodinville, Washington
- Hospital for Sick Children, Toronto, Canada
- Germany (4):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - TU Universitätsklinikum München, München
  - Fachärztin für Kinder und Jugendmedizin, Offenbach
- Israel (2):
  - HaEmek Medical Center, Afula
  - Rambam Medical Center, Haifa
- Ospedale Pediatrico Bambin Gesu - Roma, Rome, Italy
- Wakayama Medical University, Wakayama, Japan
- Kuala Lumpur Hospital, Kuala, Malaysia
- Netherlands (2):
  - Beatrix Children's Hospital, Groningen
  - Leiden University Medical, Leiden
- The Children's Memorial Health Institute, Warsaw, Poland
- Saudi Arabia (2):
  - King Fahad Medical City, Riyadh
  - Prince Sultan Riyadh Military Medical City, Riyadh
- Spain (5):
  - Germans Trias i Pujol University Hospital, Badalona
  - Hospital Sant Joan de Déu Barcelona, Esplugues de Llobregat
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clinico Universitario, Santiago de Compostela
  - Hospital Universitario Virgen del Rocio, Seville
- La Rabta Hospital, Tunis, Tunisia
- Turkey (Türkiye) (4):
  - Ihsan Dogramaci Children's Hospital, Ankara
  - Akdeniz University Hospital, Antalya
  - Çocuk Sağlığı ve Hastalıkları Anabilim Dalı, İzmit
  - Kayseri Education and Research Hospital, Kayseri
- United Kingdom (4):
  - Birmingham Children's Hospital, Birmingham
  - Royal Hospital for Sick Children, Glasgow
  - Great Ormond Street Hospital for Children, London
  - Manchester Academic Health Science Centre, Manchester